CLINICAL TRIAL: NCT04462926
Title: Evaluation of Diagnostic Accuracy of [68Ga]Ga-PSMA-11 PET/CT in Primary Staging of Intermediate and High Risk Prostatic Cancer in Men Newly Diagnosed
Acronym: PSMA-PROSTAPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Antonella Franceschetto, Prof, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ND; 2019-004685-18 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer; Prostatic Neoplasm; Urogenital Neoplasms; Prostatic Disease; Disease Attributes; Neoplasms
Keywords: 68GaPSMA PET/CT; Prostate cancer; primary staging
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms; Prostatic Diseases; Disease Attributes; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]Ga-PSMA-11 PET/CT (Experimental): 1.8-2.2 MBq (0.049-0.060 mCi) per kilogram bodyweight will be injected intravenously prior to perform the PET/CT
  Interventions: Diagnostic Test: [68Ga]Ga-PSMA-11 PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-PSMA-11 PET/CT — 1.8-2.2 MBq (0.049-0.060 mCi) per kilogram bodyweight will be injected intravenously prior to perform the PET/CT

SUMMARY:
This is a diagnostic accuracy prospective, single-centre, open-label, single group assignment interventional study.

Its aim is to evaluate the diagnostic accuracy of [68Ga]Ga-PSMA-11 PET/CT in detection of primary tumour and extra prostatic disease (lymph node, soft tissues spread or bone metastases) in men newly diagnosed with Prostate Cancer at Intermediate and High Risk, according to 2019 Prostate Cancer EAU Guidelines Risk Group Stratification (see Study Population paragraph).

The investigators are interested in the possible future role of [68Ga]Ga-labelled PSMA PET/CT as integration to conventional imaging mpMRI (with or without CT of the lower abdomen and Bone scan) in the detection of primary tumor and extra-prostatic disease (lymph node and soft tissues spread or bone metastases).

DETAILED DESCRIPTION:
This is a diagnostic accuracy prospective, single-centre, open-label, single group assignment interventional study.

The primary objective of this study is to evaluate the diagnostic accuracy of [68Ga]Ga-PSMA-11 PET/CT in detection of primary tumor and extraprostatic disease (lymph node, soft tissues spread or bone metastases) in men newly diagnosed with prostate cancer at intermediate or high-risk.

The secondary objective of this study is to compare the diagnostic accuracy of [68Ga]Ga-PSMA-11 PET/CT to the diagnostic accuracy of conventional imaging mpMRI (with or without CT of the lower abdomen and Bone scan) in the prostatic bed and extra prostatic disease in men newly diagnosed with prostate cancer at intermediate or high-risk.

To evaluate association between [68Ga]Ga-PSMA-11 PET/CT uptake value (SUVmax and SUVmean) and aggressiveness of prostate tumor (e.g. PSA serum level and Gleason Score).

ELIGIBILITY:
Inclusion Criteria:

I. Patients with histo-pathological confirmation of PCa with intermediate or high-risk disease according to 2019 Prostate Cancer EAU Guidelines Risk Group Stratification (see Study Population paragraph)

II. Patients with conventional imaging mpMRI (with or without CT of the lower abdomen and Bone scan) performed as baseline in primary PCa staging according to 2019 Prostate Cancer EAU Guidelines

III. Age >18 years/old

IV. Ability to provide written informed consent

Exclusion Criteria:

I. Contra-indication for PET/CT scan: Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam

II. Impaired renal function

III. Impaired liver function: AST or ALT > 2.5 x ULN

IV. Patients unable to understand the purpose of the study

V. Medical history of allergic reactions or hypersensitivity to [68Ga] Ga-PSMA-11 as well as to any excipient or component of the experimental medicinal product

VI. Having partecipated in clinical trial in which the experimental intervention was administered within 30 days (or 5 half-life) from administration the endovenous solution of [68Ga]Ga-PSMA-11

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy measures (sensitivity, specificity, positive and negative predictive values) of [68Ga]Ga-PSMA-11 PET/CT in detection of primary tumor and extraprostatic disease (lymph node, soft tissues spread or bone metastases). | Up to 24 months after treatment
  For the primary objective, the following index test and reference test will be considered:
  Index test: [68Ga]Ga-PSMA-11 PET/CT performed before treatment. Reference test: clinical, radiological and histo-pathologic assessment, when available, at 12 months followup and up to 24 months after treatment.
  Two nuclear medicine physicians will review the PET images using PET/CT Software Syngo.via.
  A PET positive finding for pelvic or retroperitoneal lymph nodes or lymph nodes ≥ 8mm is defined with PSMA uptake equal to or above blood pool and lower than liver.
  A PET positive finding in lymph nodes of other regions is defined with PSMA uptake equal to or above liver and lower than parotid gland. Any uptake equal to or above parotid gland will be considered positive.
  The readers will be blinded to clinical and pathologic data, except for the knowledge of diagnosis of biopsy proven prostate cancer.

SECONDARY OUTCOMES:
Comparation diagnostic accuracy of the [68Ga]Ga-PSMA-11 PET/CT versus the conventional imaging mpMRI (with or without CT of the lower abdomen and Bone scan) in the prostatic bed and extra prostatic disease. | Up to 24 months after treatment
  For the secondary objective, the following index test and reference test will be considered:
  Index test: conventional imaging mpMRI performed before treatment. Reference test: clinical, radiological and histo-pathologic assessment at 12 months follow-up and up to 24 months after treatment.
  MRI imaging results will be evaluated by two radiologists specializing in body MRI imaging with the PI-RADS version 2 criteria.
  In addition, for the secondary objective, after testing the assumption of normality with the Kolmogorov-Smirnov test, the metabolic PET parameters (SUV max and SUV mean) will be correlated with PSA serum level, by using the Pearson correlation, and with Gleason score and tumor volume, by using the Spearman correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Undecided